CLINICAL TRIAL: NCT06044168
Title: Feasibility Study: Nutritional Supplements to Support Muscle Growth in Children With Cerebral Palsy
Brief Title: Feasibility Nutritional Supplements for Muscle Growth in CP
Acronym: Nut-CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Kaat Desloovere, Prof. dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S66961
Record Dates: First submitted 2023-07-14; First posted 2023-09-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Spastic Cerebral Palsy
Keywords: Spastic Cerebral Palsy; 3D freehand ultrasound; Muscle morphology; Nutritional supplements; Leucine; Feasibility
MeSH Terms: conditions — Cerebral Palsy | interventions — Amino Acids

STUDY DESIGN:
Intervention Model Description: There will be only one group in this feasibility study. There will be no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): Receive leucine on a daily basis for 10 weeks.
  Interventions: Dietary Supplement: Dietary Supplement: Leucine

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Leucine — 150mg/kg body mass/day
  Other Names: Amino Acid

SUMMARY:
The purpose of this study is to investigate the feasibility of a 10-week plan with a nutritional supplement (leucine) and to perform pilot analyses on the effect of leucine on macroscopic muscle morphology in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the largest cause of childhood physical disability, with a prevalence of 2 to 3 per 1000 live births. While the disorder is caused by a non-progressive lesion in the developing brain, musculoskeletal alterations progress with age. The observed neuromuscular symptoms mainly involve spasticity and muscle weakness. Macroscopic lower limb muscle properties in CP, i.e. reduced muscle volume, length, anatomical cross-sectional area (CSA), and fiber CSA, have been reported, providing convincing evidence for impaired muscle growth in children with CP, already at young ages. Nutritional supplements may improve muscle strength and cause muscle hypertrophy. Within the muscle, protein synthesis depends on the availability of the branched chain amino acids (BCAA), and mainly on the presence of leucine. This stimulatory effect is thought to be primarily mediated by the upregulation of mRNA translation via enhanced signaling through the mTOR pathway. BCAA or leucine supplements have been widely used to improve muscle strength and achieve hypertrophy. In paediatric CP groups, such muscular effect of nutritional supplementation on macroscopic intrinsic muscle properties (i.e. muscle volume, anatomical CSA and muscle belly length) has not yet been studied. Therefore, a feasibility study will be carried out to investigate the feasibility of a 10-week plan with a nutritional supplement (leucine) and to perform pilot analyses on the effect of leucine on macroscopic muscle morphology in five children with cerebral palsy. This feasibility study will provide proof of concept of the administration plan of the leucine supplement and of the study design. Additionally, it will provide data for power analyses, that will be used in a future comprehensive study, investigating the effect of leucine on macroscopic muscle properties in children with cerebral palsy. To cover safety issues blood and urine sampling will be performed to objectify the patient's nutritional state and to exclude underlying disorders that would contraindicate the use of protein supplements.

ELIGIBILITY:
Inclusion Criteria:

Spastic Cerebral Palsy (diagnosed by a neuro-pediatrician from the CP Reference Centre of the University Hospital Leuven)

* Uni- of bilateral involvement
* Level II or III on the Gross Motor Function Classification System (GMFCS)
* Muscle volume for the medial gastrocnemius (target muscle) of at least 20% compared to the expected muscle volume in age-matched typically developing children

Exclusion Criteria:

* Presence of dyskinesia or ataxia
* Severe co-morbidities
* Botulinum toxin treatment ten months prior to assessment
* Previous orthopedic or neurosurgery
* Severe ankle deformities preventing fitting in test positions
* Ankle range of motion (ROM) <30% of normal values

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Patient adherence to the nutritional supplements | Between the start and the end of the 10-week nutritional plan.
  The patients adherence to the nutritional supplements will be based on data of the log book that will be used by the parents to record the time of consumption of the supplements. These data will be summarized per patient to define the number of successful nutritional supplements per week and describe the nutrition status during the period with nutritional supplements.
Overall changes in muscle volume of the medial gastrocnemius | At the start and the end of the 10-week nutritional plan
  Estimation of the muscle belly volume by 3DfUS. Muscle volume will be normalized to anthropometric growth.
Overall changes in muscle length of the medial gastrocnemius | At the start and the end of the 10-week nutritional plan
  Estimation of the muscle belly length, tendon length and muscle tendon unit complex length by 3DfUS. Muscle lengths will be normalized to anthropometric growth.
Overall changes in muscle cross-sectional area at 50% of muscle belly length | At the start and the end of the 10-week nutritional plan
  Estimation of the muscle belly cross-sectional area at 50% of the muscle belly length. Muscle cross-sectional area will be normalized to anthropometric growth.
Overall changes in echo-intensity of the medial gastrocnemius | At the start and the end of the 10-week nutritional plan
  Estimation of the echo-intensity by 3DfUS

SECONDARY OUTCOMES:
Functional strength test | At the start and the end of the 10-week nutritional plan
  Number of repetitions of bipodal toe standing possible in 30 seconds
3-day food record | Before the start of the 10-week nutritional plan
  Evaluation of the child's nutritional status, to define the amount of daily energy (kcal/kg/d) and protein (g/kg/d) intake and to estimate at which timepoint of the day the largest protein amount is consumed
Global body composition | At the start and the end of the 10-week nutritional plan
  Fat mass, fat-free mass and individual variables (e.g. resistance) will be assessed via bioelectrical impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Desloovere, Prof. dr., Principal Investigator — Department of Rehabilitation Sciences, KU Leuven, Belgium
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No